CLINICAL TRIAL: NCT06125886
Title: A Multicenter Clinical Study on Endometrial Cancer Screening in High-risk Populations in China
Brief Title: Endometrial Cancer Screening in High-risk Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Wang Jianliu, professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Endometrial cancer screening
Record Dates: First submitted 2023-10-26; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Cancer Screening
Keywords: cancer screening; endometrial cancer; endometrial atypical hyperplasia; microscale endometrial sampling; transvaginal ultrasound
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- high risk population (Experimental): The enrolled patients underwent simultaneous transvaginal ultrasound examination and microscale endometrial sampling biopsy.
  Interventions: Diagnostic Test: transvaginal ultrasound and microscale endometrial sampling biopsy

INTERVENTIONS:
Diagnostic Test: transvaginal ultrasound and microscale endometrial sampling biopsy — Transvaginal ultrasound and endometrial micro tissue pathology examination are used concurrently for endometrial cancer screening in high-risk populations. The specificity, sensitivity, and optimal combination of the two screening methods are clarified, and a cost-effectiveness analysis is conducted on different screening strategy.

SUMMARY:
Endometrial cancer is one of the most common malignancies of the reproductive system. The incidence of endometrial cancer has increased in recent years. No effective, low-cost screening method for populations at high risk exists.

The traditional methods of endometrial cancer screening and diagnosis (segmented scraping and hysteroscopic biopsy) are invasive examinations with high medical costs. It is urgent to establish a reasonable, effective, economical, and non-invasive endometrial cancer screening strategy. This study aims to evaluate the effectiveness and feasibility of transvaginal ultrasound and microscale endometrial sampling biopsy in screening for endometrial precancerous lesions and endometrial cancer among high-risk populations in China, and to conduct cost-effectiveness analysis of different screening strategy, ultimately guiding the development of screening strategies that are suitable for high-risk populations in China.

DETAILED DESCRIPTION:
The enrolled patients underwent simultaneous transvaginal ultrasound examination and microscale endometrial sampling biopsy.

After enrollment, a vaginal ultrasound examination was performed to record the thickness of the endometrium, whether there were uterine cavity masses, endometrial unevenness, and endometrial blood flow. If any of the following occurs, it is considered a positive screening result:

A. Premenopausal women with endometrial thickness greater than 8mm B. Postmenopausal endometrial thickness>4mm C. Uneven endometrium D. Abnormal echo in the uterine cavity E. Endometrium or uterine cavity with abundant blood flow (RI ≤ 0.45) If the above situation does not occur, it is considered as negative for transvaginal ultrasound screening.

After completing the transvaginal ultrasound examination, the patient used Li rush in the diagnostic room to obtain endometrial tissue samples and conduct pathological examination of the endometrial tissue.

A. Not satisfied with the specimen (mucus or hemorrhagic necrotic tissue) or insufficient sampling (only a small amount of endometrial tissue can be seen, less than 5 endometrial glands cannot be diagnosed by pathology) or no endometrial components are found, and a small amount of cervical tissue is scraped B. Normal proliferative phase, secretory phase, atrophic endometrium C. Without atypical endometrial proliferative lesions D. Suspected malignant tumor cells and tissue components E. Atypical endometrial hyperplasia/EIN or endometrial cancer If result A appears, it is considered a failure to obtain the sample, and if result B appears, it is considered a negative screening result. C. The results of D and E are considered positive for screening.

If there is a positive result in either vaginal ultrasound or endometrial microstructural pathological examination, further hysteroscopic staging and scraping of endometrial tissue pathological examination shall be performed.

follow-up

1. If the results of transvaginal ultrasound and microscale endometrial sampling biopsy are negative, a follow-up examination of transvaginal ultrasound and microscale endometrial sampling biopsy will be conducted one year later. If a positive result is found on the follow-up examination, further hysteroscopy/segmented curettage of endometrial tissue pathology will be performed.
2. Those who showed negative results on transvaginal ultrasound but failed to obtain endometrial tissue pathology examination (result A): Three months later, they underwent a follow-up examination of transvaginal ultrasound and microscale endometrial sampling biopsy. Those who showed positive results on the follow-up examination were further subjected to hysteroscopy/segmented curettage of endometrial tissue pathology examination.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 years old
2. Hypertension
3. Diabetes
4. Obesity (BMI ≥ 28)
5. History of estrogen application without progesterone antagonism
6. Polycystic ovary syndrome
7. Functional ovarian tumors (ovarian tumors that secrete estrogen) before surgical treatment
8. Infertility
9. During tamoxifen treatment, long-term use of mifepristone (greater than 3 months)
10. Abnormal uterine bleeding or vaginal discharge
11. Postmenopausal vaginal bleeding or vaginal discharge
12. Hereditary non polyposis colorectal cancer (HNPCC) patients over 35 years old, or patients with a family history of colorectal cancer or endometrial cancer
13. Cervical cytology examination indicates atypical glandular cells (AGC)
14. Previous history of ovarian cancer or breast cancer

Exclusion Criteria:

1. Body temperature ≥ 37.5 ℃
2. Acute and subacute reproductive tract inflammation
3. Suspected pregnancy
4. Clearly diagnosed patients with malignant tumors of the reproductive tract
5. Acute severe systemic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22000 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity | 2 years
  Evaluate the sensitivity and specificity of transvaginal ultrasound and endometrial microstructural pathology examination for endometrial cancer screening in high-risk populations, and determine the most effective screening mode

SECONDARY OUTCOMES:
cost-effectiveness analysis | 2 years
  Using Quality Adjusted Life Year (QALY) as the effectiveness indicator, screening expenses (screening organization management expenses, testing and evaluation expenses, personal direct expenses, and personal indirect expenses) and treatment expenses (including hospitalization expenses, outpatient expenses, direct non medical expenses, and indirect expenses) as the cost of expenditure, Calculate the cost-effectiveness ratio of different screening modes (single B-ultrasound, single endometrial micro tissue examination, B-ultrasound+endometrial micro tissue examination, B-ultrasound endometrial micro tissue examination), and calculate the cost of each extended QALY for each group and the incremental cost-effectiveness ratio between each group, and compare it with the willingness to pay value (budget line).

CONTACTS AND LOCATIONS:
Overall Officials: Jianliu Wang, doctor, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Gu B, Shang X, Yan M, Li X, Wang W, Wang Q, Zhang C. Variations in incidence and mortality rates of endometrial cancer at the global, regional, and national levels, 1990-2019. Gynecol Oncol. 2021 May;161(2):573-580. doi: 10.1016/j.ygyno.2021.01.036. Epub 2021 Feb 5. PMID 33551200
- [Background] Smith RA, von Eschenbach AC, Wender R, Levin B, Byers T, Rothenberger D, Brooks D, Creasman W, Cohen C, Runowicz C, Saslow D, Cokkinides V, Eyre H; ACS Prostate Cancer Advisory Committee, ACS Colorectal Cancer Advisory Committee, ACS Endometrial Cancer Advisory Committee. American Cancer Society guidelines for the early detection of cancer: update of early detection guidelines for prostate, colorectal, and endometrial cancers. Also: update 2001--testing for early lung cancer detection. CA Cancer J Clin. 2001 Jan-Feb;51(1):38-75; quiz 77-80. doi: 10.3322/canjclin.51.1.38. PMID 11577479
- [Background] Emons G, Steiner E, Vordermark D, Uleer C, Bock N, Paradies K, Ortmann O, Aretz S, Mallmann P, Kurzeder C, Hagen V, van Oorschot B, Hocht S, Feyer P, Egerer G, Friedrich M, Cremer W, Prott FJ, Horn LC, Prompeler H, Langrehr J, Leinung S, Beckmann MW, Kimmig R, Letsch A, Reinhardt M, Alt-Epping B, Kiesel L, Menke J, Gebhardt M, Steinke-Lange V, Rahner N, Lichtenegger W, Zeimet A, Hanf V, Weis J, Mueller M, Henscher U, Schmutzler RK, Meindl A, Hilpert F, Panke JE, Strnad V, Niehues C, Dauelsberg T, Niehoff P, Mayr D, Grab D, Kreissl M, Witteler R, Schorsch A, Mustea A, Petru E, Hubner J, Rose AD, Wight E, Tholen R, Bauerschmitz GJ, Fleisch M, Juhasz-Boess I, Sigurd L, Runnebaum I, Tempfer C, Nothacker MJ, Blodt S, Follmann M, Langer T, Raatz H, Wesselmann S, Erdogan S. Interdisciplinary Diagnosis, Therapy and Follow-up of Patients with Endometrial Cancer. Guideline (S3-Level, AWMF Registry Nummer 032/034-OL, April 2018) - Part 1 with Recommendations on the Epidemiology, Screening, Diagnosis and Hereditary Factors of Endometrial Cancer. Geburtshilfe Frauenheilkd. 2018 Oct;78(10):949-971. doi: 10.1055/a-0713-1218. Epub 2018 Oct 19. PMID 30364388
- [Background] Saccardi C, Vitagliano A, Marchetti M, Lo Turco A, Tosatto S, Palumbo M, De Lorenzo LS, Vitale SG, Scioscia M, Noventa M. Endometrial Cancer Risk Prediction According to Indication of Diagnostic Hysteroscopy in Post-Menopausal Women. Diagnostics (Basel). 2020 Apr 27;10(5):257. doi: 10.3390/diagnostics10050257. PMID 32349386
- [Background] Burnley C, Dudding N, Parker M, Parsons P, Whitaker CJ, Young W. Glandular neoplasia and borderline endocervical reporting rates before and after conversion to the SurePath(TM) liquid-based cytology (LBC) system. Diagn Cytopathol. 2011 Dec;39(12):869-74. doi: 10.1002/dc.21471. Epub 2010 Nov 2. PMID 22081523
- [Result] Matsuo K, Mandelbaum RS, Matsuzaki S, Klar M, Roman LD, Wright JD. Ovarian conservation for young women with early-stage, low-grade endometrial cancer: a 2-step schema. Am J Obstet Gynecol. 2021 Jun;224(6):574-584. doi: 10.1016/j.ajog.2020.12.1213. Epub 2021 Jan 4. PMID 33412129
- [Result] Kawaguchi R, Matsumoto K, Akira S, Ishitani K, Iwasaku K, Ueda Y, Okagaki R, Okano H, Oki T, Koga K, Kido M, Kurabayashi T, Kuribayashi Y, Sato Y, Shiina K, Takai Y, Tanimura S, Chaki O, Terauchi M, Todo Y, Noguchi Y, Nose-Ogura S, Baba T, Hirasawa A, Fujii T, Fujii T, Maruyama T, Miyagi E, Yanagida K, Yoshino O, Iwashita M, Maeda T, Minegishi T, Kobayashi H. Guidelines for office gynecology in Japan: Japan Society of Obstetrics and Gynecology (JSOG) and Japan Association of Obstetricians and Gynecologists (JAOG) 2017 edition. J Obstet Gynaecol Res. 2019 Apr;45(4):766-786. doi: 10.1111/jog.13831. Epub 2019 Jan 24. PMID 30675969
- [Result] Aue-Aungkul A, Kleebkaow P, Kietpeerakool C. Incidence and risk factors for insufficient endometrial tissue from endometrial sampling. Int J Womens Health. 2018 Aug 15;10:453-457. doi: 10.2147/IJWH.S172696. eCollection 2018. PMID 30147382
- [Result] Li MX, Zhou R, Liu C, Shen DH, Zhao LJ, Wang JL, Wei LH. Direct uterine sampling using the SAP-l sampler device to detect endometrial lesions during histopathological examination. Eur J Gynaecol Oncol. 2017;38(2):221-226. PMID 29953784
- [Result] Zhang G, Wang Y, Liang XD, Zhou R, Sun XL, Wang JL, Wei LH. Microscale endometrial sampling biopsy in detecting endometrial cancer and atypical hyperplasia in a population of 1551 women: a comparative study with hysteroscopic endometrial biopsy. Chin Med J (Engl). 2020 Sep 30;134(2):193-199. doi: 10.1097/CM9.0000000000001109. PMID 33009021